CLINICAL TRIAL: NCT03377361
Title: A Study Of Nivolumab In Combination With Trametinib With Or Without Ipilimumab In Participants With Previously Treated Metastatic Colorectal Cancers
Brief Title: An Investigational Immuno-therapy Study Of Nivolumab In Combination With Trametinib With Or Without Ipilimumab In Participants With Previously Treated Cancer of the Colon or Rectum That Has Spread
Acronym: CheckMate 9N9
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9N9; 2017-001830-24 (EudraCT Number)
Record Dates: First submitted 2017-12-14; First posted 2017-12-19 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; Colorectal Tumors; Colorectal Carcinoma; Colorectal Neoplasm
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab; trametinib; Ipilimumab; regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 Cohort 1 3rd Line (3L): nivolumab + trametinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Trametinib
- Part 1A Cohort 2 2nd Line (2L): nivolumab + ipilimumab + trametinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Trametinib; Biological: Ipilimumab
- Part 1A Cohort 3 (2L): nivolumab + ipilimumab + trametinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Trametinib; Biological: Ipilimumab
- Part 2 Cohort 4 (3L): nivolumab + ipilimumab + trametinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Trametinib; Biological: Ipilimumab
- Part 2 Cohort 5 (3L): Regorafenib (Experimental)
  Interventions: Drug: Regorafenib
- Part 1B Cohort 6 (2L): nivolumab + ipilimumab + trametinib (Experimental)
  Interventions: Biological: Nivolumab; Drug: Trametinib; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo; BMS-936558
  Arms: Part 1 Cohort 1 3rd Line (3L): nivolumab + trametinib; Part 1A Cohort 2 2nd Line (2L): nivolumab + ipilimumab + trametinib; Part 1A Cohort 3 (2L): nivolumab + ipilimumab + trametinib; Part 1B Cohort 6 (2L): nivolumab + ipilimumab + trametinib; Part 2 Cohort 4 (3L): nivolumab + ipilimumab + trametinib
Drug: Trametinib — Specified dose on specified days
  Other Names: Mekinist
  Arms: Part 1 Cohort 1 3rd Line (3L): nivolumab + trametinib; Part 1A Cohort 2 2nd Line (2L): nivolumab + ipilimumab + trametinib; Part 1A Cohort 3 (2L): nivolumab + ipilimumab + trametinib; Part 1B Cohort 6 (2L): nivolumab + ipilimumab + trametinib; Part 2 Cohort 4 (3L): nivolumab + ipilimumab + trametinib
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Part 1A Cohort 2 2nd Line (2L): nivolumab + ipilimumab + trametinib; Part 1A Cohort 3 (2L): nivolumab + ipilimumab + trametinib; Part 1B Cohort 6 (2L): nivolumab + ipilimumab + trametinib; Part 2 Cohort 4 (3L): nivolumab + ipilimumab + trametinib
Drug: Regorafenib — Specified dose on specified days
  Arms: Part 2 Cohort 5 (3L): Regorafenib

SUMMARY:
The purpose of this study is to investigate treatment with nivolumab in combination with trametinib with or without ipilimumab in participants with previously treated cancer of the colon or rectum that has spread.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed previously treated metastatic colorectal cancer with adenocarcinoma histology and in Stage IV per American Joint Committee on Cancer (version 4.0) at study entry
* Microsatellite status should be performed per local standard of practice, immunohistochemistry (IHC) and/or PCR. If IHC results are equivocal, PCR is required for determining microsatellite stable (MSS) status
* Must have measurable disease per RECIST 1.1. Participants with lesions in a previously irradiated field as the sole site of measurable disease will be permitted to enroll provided the lesion(s) have demonstrated clear progression and can be measured accurately
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 at screening and on cycle 1 day 1 (C1D1)

Exclusion Criteria:

* BRAF V600 mutant colorectal cancer
* Active brain metastases or leptomeningeal metastases
* Active, known or suspected autoimmune disease
* Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration
* History of interstitial lung disease or pneumonitis
* Prior treatment with immune checkpoint inhibitors and mitogen-activated protein kinase enzymes (MEK) inhibitors
* History of allergy or hypersensitivity to study drug components

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (47):
- United States (16):
  - Local Institution - 0022, Birmingham, Alabama
  - Local Institution - 0027, Los Angeles, California
  - Local Institution - 0067, Los Angeles, California
  - Local Institution - 0001, San Francisco, California
  - Local Institution - 0107, Gainesville, Florida
  - Local Institution - 0111, Miami, Florida
  - Local Institution - 0028, Baltimore, Maryland
  - Local Institution - 0116, Hattiesburg, Mississippi
  - Local Institution - 0103, St Louis, Missouri
  - Local Institution - 0104, New York, New York
  - Local Institution - 0029, Charlotte, North Carolina
  - Local Institution - 0100, Lancaster, Pennsylvania
  - Local Institution - 0003, Philadelphia, Pennsylvania
  - Thomas Jefferson University - Clinical Research Institute, Philadelphia, Pennsylvania
  - Local Institution - 0101, Temple, Texas
  - Local Institution - 0002, Madison, Wisconsin
- Argentina (4):
  - Local Institution - 0120, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0123, Buenos Aires, Distrito Federal
  - Local Institution - 0122, Buenos Aires, Distrito Federal
  - Local Institution - 0119, Buenos Aires
- Australia (5):
  - Local Institution - 0044, Blacktown, New South Wales
  - Local Institution - 0043, Southport, Queensland
  - Local Institution - 0068, Elizabeth Vale, South Australia
  - Local Institution - 0055, Clayton, Victoria
  - Local Institution - 0069, Heidelberg, Victoria
- Local Institution, Woluwe-Saint-Lambert, Belgium
- Canada (4):
  - Local Institution - 0113, Edmonton, Alberta
  - Local Institution - 0070, Toronto, Ontario
  - Local Institution - 0077, Montreal, Quebec
  - Local Institution - 0076, Ottawa
- Chile (2):
  - Local Institution - 0117, Santiago, Santiago Metropolitan
  - Local Institution - 0118, Santiago, Santiago Metropolitan
- Czechia (3):
  - Local Institution - 0072, Olomouc, Olomoucký kraj
  - Local Institution - 0071, Brno
  - Local Institution - 0073, Hradec Králové
- Local Institution - 0004, Hanover, Germany
- Italy (4):
  - Local Institution - 0095, Catania
  - Local Institution - 0093, Milan
  - Local Institution - 0092, Padua
  - Local Institution - 0094, Rozzano
- Spain (7):
  - Local Institution - 0079, Badalona, Barcelona [Barcelona]
  - Local Institution - 0080, Pamplona, Navarre
  - Local Institution - 0052, Barcelona
  - Local Institution - 0114, Madrid
  - Local Institution - 0051, Madrid
  - Local Institution - 0115, Madrid
  - Local Institution - 0096, Seville

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1 Cohort 1; Part 1A Cohort 2: Trame 1.5mg Cont
- Part 1 Cohort 1B: Trame 2 mg Int
- Part 1 Cohort 1D: Trame 2mg Cont
- Part 1A Cohort 2A: Trame 1mg Cont
- Part 1A Cohort 3: Trame 1.5mg Int
- Part 1A Cohort 3B: Trame 2mg Int
- Part 2 Treatment 1; Part 1B: Nivo 6 + Ipi 1 + Trame 1.5
- Part 2 Treatment 2: Regorafenib 80/160
Period: Pre-Treatment
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B | Part 2 Treatment 1 | Part 2 Treatment 2 | Part 1B
Started (Part 1 directly treated participants Part 2 randomized participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7 | 124 | 61 | 82
Completed (= Will Receive Treatment) | 3 | 3 | 6 | 7 | 3 | 3 | 7 | 121 | 57 | 82
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 0
Not completed — Subject withdrew consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Not completed — Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Period: Treatment Period
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B | Part 2 Treatment 1 | Part 2 Treatment 2 | Part 1B
Started | 3 | 3 | 6 | 7 | 3 | 3 | 7 | 121 | 57 | 82
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not Completed | 3 | 3 | 6 | 7 | 3 | 3 | 7 | 120 | 57 | 81
Not completed — Disease Progression | 3 | 2 | 5 | 3 | 3 | 3 | 6 | 106 | 48 | 59
Not completed — Study Drug Toxicity | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 2 | 16
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 3
Not completed — Adverse Event Unrelated to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 0
Not completed — Subject request to discontinue study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Subject Withdrew Consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — No longer meets study criteria | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Other Reasons | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B | Part 2 Treatment 1 | Part 2 Treatment 2 | Part 1B | Total
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7 | 124 | 61 | 82 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 3 | 5 | 6 | 2 | 3 | 6 | 89 | 47 | 60 | 223
  Between 18 and 65 years | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 35 | 14 | 22 | 76
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 0 | 4 | 2 | 1 | 3 | 48 | 30 | 37 | 129
  Male | 0 | 2 | 6 | 3 | 1 | 2 | 4 | 76 | 31 | 45 | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 10 | 6 | 7 | 25
  Not Hispanic or Latino | 3 | 3 | 6 | 6 | 3 | 2 | 7 | 55 | 27 | 51 | 163
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 59 | 28 | 24 | 111
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 5 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  White | 3 | 3 | 4 | 6 | 3 | 2 | 6 | 119 | 58 | 74 | 278
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicities in Part 1 and Part 1A
Description: Dose Limiting Toxicities are defined as adverse events have to be at least possibly related to study treatment, and not to disease progression, be clinically relevant and a clinically relevant shift from baseline.
Time Frame: 4 weeks for Doublet Reginmen and 8 weeks for triplet Regimen
Population: All treated participants in Part 1 and Part 1A
Measure: Number; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Participants | 0 | 0 | 1 | 1 | 0 | 0 | 0

2. Primary Outcome: Safety Related Events in Part 1 and Part 1 A
Description: Safety-related events in clinical trials include Adverse Events (AEs), Serious Adverse Events (SAEs), and deaths. An AE is any new or worsening medical issue in a participant receiving the study drug, regardless of its relation to the drug. This includes abnormal lab results, symptoms, or diseases. An SAE is a more severe AE that results in death, is life-threatening, requires or prolongs hospitalization, causes significant disability, involves a birth defect, or is deemed medically important-potentially jeopardizing the participant or requiring intervention, even if not immediately life-threatening. These definitions help ensure consistent reporting and evaluation of safety during clinical studies.
Time Frame: Assessed from first dose date to 100 days after last dose of study therapy. (Approximately: Part 1: ~ 6.5 Months Part 1A: ~ 5.5 Months)
Population: All treated participants in Part 1 and Part 1A
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Participants
  Adverse Events (AEs) | 3 | 3 | 6 | 7 | 3 | 3 | 7
  Drug-Related AEs | 3 | 3 | 6 | 7 | 3 | 3 | 7
  Serious Adverse Events (SAEs) | 2 | 0 | 4 | 3 | 0 | 2 | 3
  Drug-Related SAEs | 0 | 0 | 2 | 3 | 0 | 1 | 1
  Deaths | 2 | 2 | 6 | 3 | 2 | 3 | 5

3. Primary Outcome: Clinical Laboratory Abnormalities in Part 1 and Part 1A: Specific Thyroid Tests
Description: Number of participants with clinical laboratory abnormalities in specific thyroid tests
Time Frame: as for outcome 2
Population: All treated participants in Part 1 and Part 1A
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Participants
  TSH > ULN | 2 | 1 | 1 | 3 | 1 | 3 | 2
  TSH > ULN WITH TSH ≤ ULN AT BASELINE | 2 | 1 | 1 | 0 | 0 | 2 | 2
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 2 | 1 | 1 | 1 | 0 | 1 | 1
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES ≥ LLN | 0 | 0 | 0 | 2 | 1 | 2 | 1
  TSH > ULN WITH FT3/FT4 TEST MISSING | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TSH < LLN | 2 | 0 | 2 | 2 | 2 | 1 | 2
  TSH <LLN WITH TSH ≥ LLN AT BASELINE | 1 | 0 | 2 | 1 | 2 | 1 | 2
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 2 | 0 | 1 | 1 | 0 | 1 | 2
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES ≤ ULN | 0 | 0 | 1 | 0 | 2 | 0 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Clinical Laboratory Abnormalities in Part 1 and Part 1A: Specific Liver Tests
Description: Number of participants with clinical laboratory abnormalities in specific liver tests.
Time Frame: as for outcome 2
Population: All treated participants in Part 1 and Part 1A with atleast 1 On-Treatment Liver Test Measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Participants
  ALT OR AST > 3XULN | 0 | 0 | 2 | 1 | 1 | 0 | 2
  ALT OR AST> 5XULN | 0 | 0 | 2 | 1 | 1 | 0 | 2
  ALT OR AST> 10XULN | 0 | 0 | 2 | 1 | 0 | 0 | 2
  ALT OR AST > 20XULN | 0 | 0 | 1 | 1 | 0 | 0 | 0
  TOTAL BILIRUBIN > 2XULN | 0 | 0 | 2 | 0 | 0 | 0 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0 | 0 | 2 | 0 | 0 | 0 | 1
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0 | 0 | 2 | 0 | 0 | 0 | 1

5. Primary Outcome: Overal Response Rate in Part 1B and Part 2
Description: ORR is defined as the proportion of all treated participants whose BOR is either confirmed complete response (CR) or confirmed partial response (PR).
Time Frame: Approximately up to 30 Months
Population: All Randomized Participants in Part 1B and Part 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1B | Part 2 Treatment 1 | Part 2 Treatment 2
Number analyzed (Participants) | 82 | 124 | 61
Percentage of Participants | 9.8 [4.3 to 18.3] | 1.6 [0.2 to 5.7] | 1.6 [0.0 to 8.8]

6. Secondary Outcome: Objective Response Rate in Part 1 and Part 1A
Description: as for outcome 5
Time Frame: From the first dosing date and the date of the initial objectively documented tumor progression or subsequent therapy date (Approximately up to 21 Months)
Population: All treated participants in Part 1 and Part 1A
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Percentage of Participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 45.9] | 28.6 [3.7 to 71.0] | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0]

7. Secondary Outcome: Disease Control Rate in Part 1 and Part 1A
Description: The disease control rate (DCR) is defined as the percentage of participants whose BOR is either confirmed CR or confirmed PR or stable disease (SD)
Time Frame: as for outcome 6
Population: All treated participants in Part 1 and Part 1A
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Percentage of Participants | 66.7 [9.4 to 99.2] | 33.3 [0.8 to 90.6] | 50.0 [11.8 to 88.2] | 57.1 [18.4 to 90.1] | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 28.6 [3.7 to 71.0]

8. Secondary Outcome: Duration of Response in Part 1 and Part 1A
Description: DOR for a participant with a BOR of confirmed CR or PR, is defined as the time between the date of first confirmed response and the date of the first objectively documented tumor progression per RECIST 1.1 or death, whichever occurs first.
Time Frame: Approximately up to 20 Months
Population: All treated participants in Part 1 and Part 1A who had a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Months |  |  |  | 9.46 [NA to NA] — Insufficient number of events to calculate via KM Methodology. | 19.42 [NA to NA] — Insufficient number of events to calculate via KM methodology. |  |

9. Secondary Outcome: Time to Response in Part 1 and Part 1A
Description: Time to response (TTR) is defined for participants who had a confirmed CR or PR as the time from the first dosing date to the date of first documented CR or PR per RECIST 1.1.
Time Frame: From the first dosing date to the date of first documented CR or PR per RECIST 1.1. (Approximately on average 10 months)
Population: All treated participants in Part 1 and Part 1A who had a response
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 0 | 0
Months |  |  |  | 5.63 [1.8 to 9.5] | 1.54 [1.54 to 1.54] |  |

10. Secondary Outcome: Progression Free Survival in Part 1 and Part 1A
Description: PFS for a participant is defined as the time from the first dosing date to the date of first objectively documented disease progression per RECIST 1.1 (ie, radiologic) or death due to any cause, whichever occurs first.
Time Frame: from the first dosing date to the date of first objectively documented disease progression or death, whichever occurs first (Approximately up to 21 months)
Population: All treated participants in Part 1 and Part 1A
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Months | 3.58 [1.84 to NA] — Insufficient number of participants with events to calculate via KM methodology | 1.91 [1.74 to NA] — Insufficient number of participants with events to calculate via KM methodology | 2.66 [0.79 to NA] — Insufficient number of participants with events to calculate via KM methodology | 7.36 [1.84 to NA] — Insufficient number of participants with events to calculate via KM methodology | 1.74 [1.74 to NA] — Insufficient number of participants with events to calculate via KM methodology | 4.14 [1.84 to NA] — Insufficient number of participants with events to calculate via KM methodology | 1.81 [0.92 to NA] — Insufficient number of participants with events to calculate via KM methodology

11. Secondary Outcome: Overall Survival in Part 1 and Part 1A
Description: OS for a participant is defined as the time from the first dosing date to the date of death due to any cause. A participant who has not died will be censored at last known date alive.
Time Frame: Approximately up to 69 Months
Population: All treated participants in Part 1 and Part 1A
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B
Number analyzed (Participants) | 3 | 3 | 6 | 7 | 3 | 3 | 7
Months | 8.99 [8.80 to NA] — Insufficient number of participants with events to calculate via KM methodology | 18.50 [17.45 to NA] — Insufficient number of participants with events to calculate via KM methodology | 9.61 [0.89 to NA] — Insufficient number of participants with events to calculate via KM methodology | 42.09 [11.60 to NA] — Insufficient number of participants with events to calculate via KM methodology | 19.02 [8.80 to NA] — Insufficient number of participants with events to calculate via KM methodology | 11.33 [10.51 to NA] — Insufficient number of participants with events to calculate via KM methodology | 36.24 [2.23 to NA] — Insufficient number of participants with events to calculate via KM methodology

12. Secondary Outcome: Safety Related Events in Part 1B and Part 2
Description: as for outcome 2
Time Frame: Assessed from first dose date to 100 days after last dose of study therapy. (Approximately: 6.8 Months)
Population: All Treated Participants in Part 1B and Part 2
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B | Part 2 Treatment 1 | Part 2 Treatment 2
Number analyzed (Participants) | 82 | 121 | 57
Participants
  Adverse Events (AEs) | 82 | 121 | 57
  Drug-Related AEs | 80 | 116 | 52
  Serious Adverse Events (SAEs) | 36 | 56 | 19
  Drug-Related SAEs | 20 | 21 | 3
  Deaths | 49 | 106 | 53

13. Secondary Outcome: Clinical Laboratory Abnormalities in Part 1B and Part 2: Specific Thyroid Tests
Description: Number of participants with clinical laboratory abnormalities in specific thyroid tests
Time Frame: Assessed from first dose date to 100 days after last dose of study therapy. (Approximately: 6.8 Months)
Population: All Treated Participants in Part 1B and Part 2 with atleast 1 On-Treatment TSH Measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B | Part 2 Treatment 1 | Part 2 Treatment 2
Number analyzed (Participants) | 81 | 114 | 46
Participants
  TSH > ULN | 13 | 31 | 21
  TSH > ULN WITH TSH ≤ ULN AT BASELINE | 9 | 18 | 16
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 9 | 14 | 3
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES ≥ LLN | 3 | 13 | 14
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1 | 4 | 4
  TSH < LLN | 14 | 24 | 0
  TSH <LLN WITH TSH ≥ LLN AT BASELINE | 11 | 21 | 0
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 5 | 12 | 0
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES ≤ ULN | 8 | 7 | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 1 | 5 | 0

14. Secondary Outcome: Clinical Laboratory Abnormalities in Part 1B and Part 2: Specific Liver Tests
Description: Number of participants with clinical laboratory abnormalities in specific liver tests.
Time Frame: Assessed from first dose date to 100 days after last dose of study therapy. (Approximately: 6.8 Months)
Population: All Treated Participants in Part 1B and Part 2 with atleast 1 On-Treatment Liver test Measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1B | Part 2 Treatment 1 | Part 2 Treatment 2
Number analyzed (Participants) | 82 | 121 | 57
Participants
  ALT OR AST > 3XULN | 18 | 38 | 11
  ALT OR AST> 5XULN | 8 | 19 | 8
  ALT OR AST> 10XULN | 1 | 5 | 4
  ALT OR AST > 20XULN | 0 | 3 | 2
  TOTAL BILIRUBIN > 2XULN | 3 | 9 | 12
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 2 | 6 | 7
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 2 | 7 | 7

ADVERSE EVENTS:
Time Frame: Part 1: Approximately 5.5 Months Part 1A: Approximately 6.5 Months Part 1B and 2: Approximately 6.8 Months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- Part 1 Cohort 1; Part 1A Cohort 2: Trame 1.5 mg Cont
- Part 1 Cohort 1D: Trame 2 mg Cont
- Part 1A Cohort 2A: Trame 1 mg Cont
- Part 1A Cohort 3: Trame 1.5 mg Int
- Part 1A Cohort 3B: Trame 2 mg Int
Arm/Group | Part 1 Cohort 1 | Part 1 Cohort 1B | Part 1 Cohort 1D | Part 1A Cohort 2 | Part 1A Cohort 2A | Part 1A Cohort 3 | Part 1A Cohort 3B | Part 1B | Part 2 Treatment 1 | Part 2 Treatment 2
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 6/6 | 3/7 | 2/3 | 3/3 | 5/7 | 49/82 | 108/124 | 55/61
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 5/6 | 3/7 | 0/3 | 2/3 | 3/7 | 42/82 | 79/121 | 33/57
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 7/7 | 3/3 | 3/3 | 7/7 | 82/82 | 121/121 | 55/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=3) | Part 1 Cohort 1B (N=3) | Part 1 Cohort 1D (N=6) | Part 1A Cohort 2 (N=7) | Part 1A Cohort 2A (N=3) | Part 1A Cohort 3 (N=3) | Part 1A Cohort 3B (N=7) | Part 1B (N=82) | Part 2 Treatment 1 (N=121) | Part 2 Treatment 2 (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Detachment of retinal pigment epithelium (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 3 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Gastrooesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac death (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 5 | 7 | 2
Acute cholecystitis necrotic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary cast syndrome (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Listeriosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Pneumonia pneumococcal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proteus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood lactic acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 42 | 21
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to eye (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extrinsic iliac vein compression (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1 Cohort 1 (N=3) | Part 1 Cohort 1B (N=3) | Part 1 Cohort 1D (N=6) | Part 1A Cohort 2 (N=7) | Part 1A Cohort 2A (N=3) | Part 1A Cohort 3 (N=3) | Part 1A Cohort 3B (N=7) | Part 1B (N=82) | Part 2 Treatment 1 (N=121) | Part 2 Treatment 2 (N=57)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 4 | 1 | 2 | 4 | 18 | 36 | 12
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 4 | 6
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 3 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4 | 2 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 7 | 4 | 2
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 5 | 2 | 0
Iridocyclitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Subretinal fluid (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Swelling of eyelid (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2 | 1 | 1 | 18 | 17 | 9
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 5 | 4
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 7 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 1 | 1 | 2 | 10 | 17 | 13
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 4 | 6 | 2 | 2 | 4 | 45 | 52 | 22
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 6 | 7 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 7 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 2 | 5 | 1 | 2 | 5 | 26 | 55 | 9
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 7 | 10 | 8
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 2 | 2 | 2 | 2 | 17 | 36 | 5
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 31 | 16
Chills (General disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 4 | 9 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 4 | 7 | 3 | 1 | 6 | 33 | 51 | 22
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 2 | 0
Malaise (General disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 7 | 7 | 9
Oedema peripheral (General disorders) | 2 | 1 | 3 | 0 | 1 | 1 | 1 | 7 | 31 | 3
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 3 | 17 | 28 | 13
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 9 | 4
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 5 | 5 | 3
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 6 | 6
Candida infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 3 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 7 | 2
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 4 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 14 | 28 | 13
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 20 | 37 | 17
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 13 | 6
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 5 | 10 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 16 | 19
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 5 | 8 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 6 | 3
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4 | 6
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 10 | 4
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 8 | 7
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Weight decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 6 | 17 | 10
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 4 | 2 | 2 | 1 | 1 | 13 | 32 | 15
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 5 | 11 | 10
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 0 | 1 | 1 | 5 | 9 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 2 | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 5 | 12 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 6 | 9 | 8
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 9 | 11 | 4
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 6 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 6 | 5
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 0 | 0 | 2 | 8 | 6 | 2
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 10 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 13 | 8 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 11 | 5
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4 | 4 | 5
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 1 | 5 | 14 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 5 | 23 | 5
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 8 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 3 | 5 | 4 | 3 | 3 | 6 | 20 | 39 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 9 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 25
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 3 | 27 | 31 | 5
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 4 | 0 | 0 | 3 | 39 | 51 | 6
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 16 | 13 | 6
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 13 | 10 | 7
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/61/NCT03377361/Prot_SAP_000.pdf